CLINICAL TRIAL: NCT05018013
Title: Efficacy and Safety of Ammoxetine Hydrochloride Enteric-coated Tablets in Subjects With Depression: A Multicenter, Randomized, Double-blind, Double-dummy, Active- and Placebo-controlled, Parallel-group, Phase II Study
Brief Title: Study of Ammoxetine Hydrochloride Enteric-coated Tablets in Subjects With Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HA1406-CSP-003
Record Dates: First submitted 2021-07-30; First posted 2021-08-24 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ammoxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Duloxetine group (Active Comparator): The eligible subjects will receive duloxetine hydrochloride enteric-coated capsules plus placebo to Ammoxetine.
  Interventions: Drug: Duloxetine hydrochloride enteric-coated capsules; Drug: Placebo to Ammoxetine
- Placebo group (Placebo Comparator): The eligible subjects will receive placebo to Ammoxetine and placebo to Duloxetine.
  Interventions: Drug: Placebo to Ammoxetine; Drug: Placebo to Duloxetine
- Ammoxetine group-cohort 1 (Experimental): The eligible subjects will receive Ammoxetine hydrochloride enteric-coated tablets plus placebo to Duloxetine.
  Interventions: Drug: Ammoxetine hydrochloride enteric-coated tablets; Drug: Placebo to Duloxetine
- Ammoxetine group-cohort 2 (Experimental): The eligible subjects will receive Ammoxetine hydrochloride enteric-coated tablets plus placebo to Duloxetine.
  Interventions: Drug: Ammoxetine hydrochloride enteric-coated tablets; Drug: Placebo to Duloxetine
- Ammoxetine group-cohort 3 (Experimental): The eligible subjects will receive Ammoxetine hydrochloride enteric-coated tablets plus placebo to Duloxetine.
  Interventions: Drug: Ammoxetine hydrochloride enteric-coated tablets; Drug: Placebo to Duloxetine
- Ammoxetine group-cohort 4 (Experimental): The eligible subjects will receive Ammoxetine hydrochloride enteric-coated tablets plus placebo to Duloxetine.
  Interventions: Drug: Ammoxetine hydrochloride enteric-coated tablets; Drug: Placebo to Duloxetine

INTERVENTIONS:
Drug: Ammoxetine hydrochloride enteric-coated tablets — Ammoxetine hydrochloride enteric-coated tablets
  Other Names: Ammoxetine
  Arms: Ammoxetine group-cohort 1; Ammoxetine group-cohort 2; Ammoxetine group-cohort 3; Ammoxetine group-cohort 4
Drug: Duloxetine hydrochloride enteric-coated capsules — Duloxetine hydrochloride enteric-coated capsules
  Other Names: Duloxetine
  Arms: Duloxetine group
Drug: Placebo to Ammoxetine — Placebo to Ammoxetine
  Other Names: Placebo
  Arms: Duloxetine group; Placebo group
Drug: Placebo to Duloxetine — Placebo to Duloxetine
  Other Names: Placebo
  Arms: Ammoxetine group-cohort 1; Ammoxetine group-cohort 2; Ammoxetine group-cohort 3; Ammoxetine group-cohort 4; Placebo group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ammoxetine hydrochloride enteric-coated tablets in subjects with depression.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, duloxetine hydrochloride enteric coated capsule positive and placebo-controlled multicenter study was used to evaluate the efficacy and safety of different doses of amxetine hydrochloride enteric coated tablets in the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects aged 18 and 65 years (inclusive), no gender limitation;
* 2. Subject has recurrent Major Depressive Disorder (MDD) as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5, 5th Edition), single episode or recurrent episodes (DSM-IV-TR criteria, classification code 296.2/296.3), without psychotic symptoms;
* 3. Subjects with a Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 26 and subjects with Clinical Global Impression Scale Disease Severity CGI-S severity score ≥ 4 at screening and baseline;
* 4. For male or female with fertility: must agree to use effective contraceptive method during the study and within 1 month after the end of the trial;
* 5. Be able to read and understand the content of the informed consent and voluntarily sign the informed consent.

Exclusion Criteria:

* 1. Subjects with ≥ 25% reduction in MADRS score in the baseline period compared to the screening period;
* 2. Subjects meet DSM-5 diagnostic criteria for other mental disorders (schizophrenia spectrum and other psychiatric disorders, bipolar and related disorders, anxiety disorders, obsessive-compulsive and related disorders, somatic symptoms and related disorders, etc.);
* 3. Subjects are diagnosed as DSM-5 drug use disorder;
* 4. Refractory depression (subjects who had previously used two different mechanisms of antidepressants and failed after receiving adequate treatment (at least 8 weeks);
* 5. Organic mental disorders, such as depression caused by hypothyroidism;
* 6. Depression caused by psychoactive substances or non-addictive substances;
* 7. Subjects with other diseases or other types of mental disorders with depressive symptoms;
* 8. Subjects assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) and those judged by the investigator to be at risk for suicide, or to have engaged in suicidal behaviour within 6 months prior to screening;
* 9. Allergic constitution (e.g. allergic to two or more drugs or to serotonin norepinephrine reuptake inhibitors (SNRIs));
* 10.Previous history of malignant tumor;
* 11.Previous history of elevated intraocular pressure or narrow angle glaucoma;
* 12.Subjects suffered from other serious physical diseases, such as uncontrolled hypertension or unstable cardiovascular disease, serious liver disease, kidney disease, blood disease, endocrine disease, neurological disease, etc;
* 13.Subjects with diseases that interfere with the absorption of oral medications, such as active bowel disease, partial or complete intestinal obstruction, chronic diarrhea, etc;
* 14.Subjects who have used drugs or foods that alter the activity of liver enzymes (CYP2C19 and CYP3A4) such as dexamethasone, rifampicin, omeprazole, grapefruit, etc., within 4 weeks prior to screening;
* 15.12-lead ECG system showed degree II or III atrioventricular block, long QT syndrome or QTc > 450 ms (male) / 470 ms (female) at screening;
* 16.Subjects discontinued use of a combination of drugs that prolong the QT interval prior to randomization, or drugs that can cause prolongation of the QT and may induce TdP for less than 5 half-lives of the drugs;
* 17.In screening period, subjects with ALT or AST 1.5 times higher than the upper limit of laboratory normal value; creatinine 1.1 times higher than the upper limit of normal value; and abnormalities in 2 or more of the 5 indicators of thyroid function (TSH, FT3, FT4, TT3 or TT4 0.9 times below the lower limit of normal value or 1.1 times above the upper limit of normal value);
* 18.Subjects have used monoamine oxidase inhibitors within 2 weeks before randomization;
* 19.Subjects discontinuing antipsychotics, antidepressants or mood stabilizers for less than 5 half-lives of the drug before randomization;
* 20.Subjects who are using long half-life drugs (such as fluoxetine, long-acting antipsychotics, etc.);
* 21.Subjects who have received electroconvulsive therapy (ECT), systematic psychotherapy (interpersonal relationship therapy, dynamic therapy, cognitive behavior therapy, etc.), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), phototherapy, etc. within 3 months before screening, or subjects who, in the judgment of the investigator, are currently in need of such treatment;
* 22.Female subjects who are breastfeeding or have a positive pregnancy test during the screening period or during the study;
* 23.Alcohol or drug dependence within 3 months before screening;
* 24.Subjects who have participated in other clinical trials within 3 months before screening and are taking the test drug;
* 25.Subjects who, in the opinion of the investigator, have any other condition that makes them unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-08-21 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montgomery Asperger Depression Scale (MADRS) score at the end of treatment (week 6) | Baseline and week 6
  The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
  Change = (Week 6 post-dose score - baseline week 0 score). at the end of treatment (week 6)

SECONDARY OUTCOMES:
Change from baseline in Hamilton Depression Scale (HAMD-17) at week 1, 2, 4, 6 | Baseline, week 1, 2, 4 and 6
  The HAMD-17 is a 17-item, clinician-rated scale that assesses depressive symptoms. The HAMD-17 consists of 17 symptoms, each of which is rated from 0 to 2 or 0 to 4, where 0 is none/absent. The HAMD-17 total score is calculated as the sum of the 17 individual symptom scores; the total score can range from 0 to 52. Higher HAMD-17 scores indicate more severe depression.
  Change = (Week 1, 2, 4 and 6 post-dose score - baseline week 0 score).
Change from baseline in Hamilton Anxiety Inventory (HAMA) scores at week 1, 2, 4, 6 | Baseline, week 1, 2, 4 and 6
  The HAMA is used as a rating measure of anxiety severity. The scale consists of 14 items. Each item is rated on a scale of 0 to 4. The HAMA total score is the sum of the 14 items and the score ranges from 0 to 56, 0 is considered the best outcome.
  Change = (Week 1, 2, 4 and 6 post-dose score - baseline week 0 score).
Change from baseline in CGI-S score at week 1, 2, 4, 6,7 | Baseline, week 1, 2, 4, 6 and 7
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment. The CGI-S will provide an overall clinician-determined summary measure that takes into account all available information including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function.
  Change = (Week 1, 2, 4, 6 and 7 post-dose score - baseline week 0 score).
The percentage of subjects with a MARDS score reduction ≥ 25% | Week 1 and 2
  The score reduction rate is defined as (screening period MARDS scale score - post-dose MARDS scale score)/screening period MARDS scale score x 100%.
Incidence of adverse events (AE) | Throughout the study period,an average of 18 months
  The AEs will be assessed according to the National Cancer Institute (NCI) CTCAE v5.0.
Change from baseline in MADRS score at week 1, 2, 4 | baseline, week 1, 2 and 4
  Change = (Week 1, 2 and 4 post-dose score - baseline week 0 score).

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yanli, MD, Study Director — CSPC Zhongqi Pharmaceutical Technology (Shijiazhuang) Co., Ltd; Li Huafang, Ph.D, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No